CLINICAL TRIAL: NCT06363747
Title: The Medically Reproducing Bariatric Surgery (MRB) II Study: SEMAGLUTIDE Followed by OPTIFAST in Veterans With Type 2 Diabetes
Brief Title: The Medically Reproducing Bariatric Surgery (MRB) II Study
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Optifast; Type 2 diabetes; Semglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: Control--[GLP-1 agonist +/- DM2 meds + medical management + nutritional/behavioral counseling] Experimental---[Optifast + GLP-1 agonist + medical management + nutritional/behavioral counseling]
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): Patients in the control group will attend four in-person visits with the study coordinator at baseline, week 12, week 24, and week 48 to measure study outcomes.
  Patients will get medical drug management (endocrinologist), nutritional/behavioral counseling (dietician, psychologist) and will be maintained on once weekly GLP-1 agonist +/- other diabetic medicines.
- Very Low Calorie Diet (Experimental): Patients in the experimental group will attend 4 in-person visits with the study coordinator at baseline, week 12, week 24, and week 48 to measure study outcomes. Additionally, they will undergo a 2 week run-in phase before baseline with weekly meetings to ensure that they are able to tolerate and comply with Optifast.
  Patients will get medical drug management (endocrinologist), nutritional/behavioral counseling (dietician, psychologist) and will be maintained on Optifast + once weekly GLP-1 agonist +/- other diabetic medicines.
  Interventions: Other: Very Low Calorie Diet

INTERVENTIONS:
Other: Very Low Calorie Diet — Optifast is a medically supervised very low-calorie diet (VLCD) diet that safely induces caloric restriction
  Other Names: Optifast
  Arms: Very Low Calorie Diet

SUMMARY:
Roux-en-Y (RYGB) gastric bypass reduces the size and capacity of the stomach and bypasses a portion of the small intestine which leads to decreased food intake and higher levels of a gut hormone called GLP-1 (glucagon-like-peptide-1). These changes lead to weight loss, improved blood sugars and often remission of type 2 diabetes but most patients do not qualify or want surgery. The investigators are searching for ways to make the beneficial effects of RYGB available to most type 2 diabetes patients rather than a select few that undergo RYGB.

The investigators believe that parts of RYGB can be medically reproduced through a combination of diet and medicine. Once weekly injectable GLP-1 medicine that leads to weight loss and improved blood sugar control in type 2 diabetes are now FDA approved. Optifast is a medically supervised diet that safely reduces calorie intake to 800 calories per day for three months by replacing normal meals with specially prepared bars and shakes which leads to weight loss and improved blood sugar control in type 2 diabetes. Normal meals are then gradually reintroduced over 6 weeks and the bars/shakes are stopped. The investigators hypothesize that Optifast (diet) + once weekly GLP-1 will lead to weight loss and improvement in blood sugar control in type 2 diabetes similar to what is seen after RYGB.

DETAILED DESCRIPTION:
MRB II is a two arm 50-week study that will recruit Veteran DM2 patients already on a stable dose of a GLP-1 agonist +/- DM2 agents. The investigators will recruit 50 patients and assign 25 subjects to the control arm and 25 subjects to the experimental arm. The control and experimental arm (n=25) will have in-person visits with the study PI, certified diabetes educator (CDE) and behavioral psychologist (Psych) at baseline, week 12, week 24 and week 48 to optimize glycemic control. Visits with the PI will be one-on-one but visits with CDE/Psych will be shared-medical appointments. Furthermore, the experimental arm (n=25) will also be enrolled in the Optifast medical weight loss program starting with a 2-week run-in phase to determine if they are able to tolerate Isocaloric Optifast (7 meal replacements/day) while also minimizing significant weight loss prior to the start of the study. The patients in the experimental arm successfully completing the run-in phase will then continue and enter the 50-week study.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 25-75 years
* BMI >27
* diagnosis of type 2 diabetes
* weight stable for 1 month
* hemoglobin A1C >7.0%
* on stable dose of once weekly GLP-1 agonist
* on oral or injectable DM2 medicines
* interested in losing weight
* agreeable to regular visits per study protocol
* access to telephone and reliable transportation and has a VAMC provider
* using a Freestyle Libre glucose monitoring device and/or glucometer device

Exclusion Criteria:

* age >75,
* A1C <7%
* pregnant
* breast feeding
* prior history of pancreatitis
* prior history of gastroparesis
* history of thyroid cancer/multiple endocrine neoplasia/thyroid nodules/medullary thyroid cancer (contraindication to Liraglutide)
* history of gallstones
* history of hyperoxaluria or calcium oxalate nephrolithiasis
* history of Roux-en-Y gastric bypass or gastric sleeve or any other bariatric procedure,
* type 1 diabetes
* any abnormality on the screening EKG that could subject patient to increased risk during the study
* any gastrointestinal condition causing malabsorption (including but not limited to inflammatory bowel disease, celiac sprue)
* unwilling or unable to complete scheduled testing
* any serious and/or unstable medical, psychiatric, or other condition(s) that prevents the patient from providing informed consent or complying with the study
* organ transplantation or those on immunosuppressants
* chronic anticoagulation
* recent myocardial infarction, unstable angina, stroke, coronary artery bypass or transient ischemia attacks in the past 6 months
* chronic prednisone use
* hepatitis
* cirrhosis
* GFR <50
* deep vein thrombosis in past 6 months
* active malignancy
* unstable psychiatric condition including active or current suicidal ideation
* enrolled in another research study related to diet and/or physical activity

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control | baseline, week 12, week 24, week 48
  Hemoglobin A1C

SECONDARY OUTCOMES:
Weight lost | baseline, week 12, week 24, week 48
  Percentage of weight loss
Medication Intensity | baseline, week 12, week 24, week 48
  Medication Effect Score (MES) measures the intensity of antiglycemic medicines used to treat type 2 diabetes with higher scores indicating greater medication intensity.
Health Related Quality of Life | baseline, week 12, week 24, week 48
  Problem Areas In Diabetes (PAID) is a self-administered 20-item scale. Each item is scored from 0 (not a problem) to 4 (serious problem). The sum of all item scores multiplied by 1.25 gives the total PAID score, which ranges from 0 to 100, higher scores reflecting greater emotional distress. A score of 40 or above is indicative of severe emotional distress.

OTHER OUTCOMES:
Symptom Item Checklist | 2 week run-in phase
  SCL-90-R is a self-report instrument containing 90 items and designed to measure nine current psychiatric symptoms, as well as psychological distress. The SCL-90-R sub-scales assess followings psychiatric symptoms: Somatization, Obsessive Compulsive Disorder, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism. Each item has five following response categories: 0 = Not at all, 1= little, 2 = some, 3 = very, 4 = severe.

CONTACTS AND LOCATIONS:
Overall Officials: Moahad Dar, MD, Principal Investigator — Department of Veteran Affairs
Locations (1):
- Greenville VA Health Care Center, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and/or specimens will be transported BETWEEN sites that are under the auspices of the Durham VA Medical Center. The Greenville VA Health Care Center is the primary study site. Data analysis will be conducted by HSRD located at the Durham VA medical center. Data and/or specimens will be transported to non-VA/VHA sites (e.g., academic affiliates, laboratories, etc.) as coded data which will be shared via email using Azure RMS encryption. The study will use a VA issued laptop. Direct identifiers will be maintained separately from data and or specimens by using a code to "identify" subjects. In a separate database (i.e., a "linking" or "cross-walk" database) this code will be linked to identifying subject information. Reporting of results, such as in scientific papers and presentations, will never identify individual subjects. Data will be presented in aggregate and individual-level data will not be published. No future use of data is currently planned.
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol was shared with study sponsor prior to IRB submission. Study sponsor will receive a summary of study results at study conclusion but will not have access to individually identifiable information.

REFERENCES:
- [Background] Andreadis P, Karagiannis T, Malandris K, Avgerinos I, Liakos A, Manolopoulos A, Bekiari E, Matthews DR, Tsapas A. Semaglutide for type 2 diabetes mellitus: A systematic review and meta-analysis. Diabetes Obes Metab. 2018 Sep;20(9):2255-2263. doi: 10.1111/dom.13361. Epub 2018 Jun 10. PMID 29756388
- [Background] Ard JD, Lewis KH, Rothberg A, Auriemma A, Coburn SL, Cohen SS, Loper J, Matarese L, Pories WJ, Periman S. Effectiveness of a Total Meal Replacement Program (OPTIFAST Program) on Weight Loss: Results from the OPTIWIN Study. Obesity (Silver Spring). 2019 Jan;27(1):22-29. doi: 10.1002/oby.22303. Epub 2018 Nov 13. PMID 30421863
- [Background] Bianciardi E, Gentileschi P, Niolu C, Innamorati M, Fabbricatore M, Contini LM, Procenesi L, Siracusano A, Imperatori C. Assessing psychopathology in bariatric surgery candidates: discriminant validity of the SCL-90-R and SCL-K-9 in a large sample of patients. Eat Weight Disord. 2021 Oct;26(7):2211-2218. doi: 10.1007/s40519-020-01068-2. Epub 2020 Nov 23. PMID 33226607
- [Background] Chaudhry ZW, Doshi RS, Mehta AK, Jacobs DK, Vakil RM, Lee CJ, Bleich SN, Kalyani RR, Clark JM, Gudzune KA. A systematic review of commercial weight loss programmes' effect on glycemic outcomes among overweight and obese adults with and without type 2 diabetes mellitus. Obes Rev. 2016 Aug;17(8):758-69. doi: 10.1111/obr.12423. Epub 2016 May 26. PMID 27230990
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Dar MS, Chapman WH 3rd, Pender JR, Drake AJ 3rd, O'Brien K, Tanenberg RJ, Dohm GL, Pories WJ. GLP-1 response to a mixed meal: what happens 10 years after Roux-en-Y gastric bypass (RYGB)? Obes Surg. 2012 Jul;22(7):1077-83. doi: 10.1007/s11695-012-0624-1. PMID 22419108
- [Background] Diamant M, Nauck MA, Shaginian R, Malone JK, Cleall S, Reaney M, de Vries D, Hoogwerf BJ, MacConell L, Wolffenbuttel BH; 4B Study Group. Glucagon-like peptide 1 receptor agonist or bolus insulin with optimized basal insulin in type 2 diabetes. Diabetes Care. 2014 Oct;37(10):2763-73. doi: 10.2337/dc14-0876. Epub 2014 Jul 10. PMID 25011946
- [Background] Engelgau MM, Geiss LS, Saaddine JB, Boyle JP, Benjamin SM, Gregg EW, Tierney EF, Rios-Burrows N, Mokdad AH, Ford ES, Imperatore G, Narayan KM. The evolving diabetes burden in the United States. Ann Intern Med. 2004 Jun 1;140(11):945-50. doi: 10.7326/0003-4819-140-11-200406010-00035. PMID 15172919
- [Background] Flegal KM, Carroll MD, Ogden CL, Curtin LR. Prevalence and trends in obesity among US adults, 1999-2008. JAMA. 2010 Jan 20;303(3):235-41. doi: 10.1001/jama.2009.2014. Epub 2010 Jan 13. PMID 20071471
- [Background] Henry RR, Scheaffer L, Olefsky JM. Glycemic effects of intensive caloric restriction and isocaloric refeeding in noninsulin-dependent diabetes mellitus. J Clin Endocrinol Metab. 1985 Nov;61(5):917-25. doi: 10.1210/jcem-61-5-917. PMID 4044780
- [Background] Jackness C, Karmally W, Febres G, Conwell IM, Ahmed L, Bessler M, McMahon DJ, Korner J. Very low-calorie diet mimics the early beneficial effect of Roux-en-Y gastric bypass on insulin sensitivity and beta-cell Function in type 2 diabetic patients. Diabetes. 2013 Sep;62(9):3027-32. doi: 10.2337/db12-1762. Epub 2013 Apr 22. PMID 23610060
- [Background] Kirschner MA, Schneider G, Ertel NH, Gorman J. An eight-year experience with a very-low-calorie formula diet for control of major obesity. Int J Obes. 1988;12(1):69-80. PMID 3360564
- [Background] Lingvay I, Guth E, Islam A, Livingston E. Rapid improvement in diabetes after gastric bypass surgery: is it the diet or surgery? Diabetes Care. 2013 Sep;36(9):2741-7. doi: 10.2337/dc12-2316. Epub 2013 Mar 25. PMID 23530013
- [Background] Maney M, Tseng CL, Safford MM, Miller DR, Pogach LM. Impact of self-reported patient characteristics upon assessment of glycemic control in the Veterans Health Administration. Diabetes Care. 2007 Feb;30(2):245-51. doi: 10.2337/dc06-0771. PMID 17259489
- [Background] Mann DM, Woodward M, Ye F, Krousel-Wood M, Muntner P. Trends in medication use among US adults with diabetes mellitus: glycemic control at the expense of controlling cardiovascular risk factors. Arch Intern Med. 2009 Oct 12;169(18):1718-20. doi: 10.1001/archinternmed.2009.296. No abstract available. PMID 19822830
- [Background] Mayer SB, Jeffreys AS, Olsen MK, McDuffie JR, Feinglos MN, Yancy WS Jr. Two diets with different haemoglobin A1c and antiglycaemic medication effects despite similar weight loss in type 2 diabetes. Diabetes Obes Metab. 2014 Jan;16(1):90-3. doi: 10.1111/dom.12191. Epub 2013 Aug 29. PMID 23911112
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Leccesi L, Nanni G, Pomp A, Castagneto M, Ghirlanda G, Rubino F. Bariatric surgery versus conventional medical therapy for type 2 diabetes. N Engl J Med. 2012 Apr 26;366(17):1577-85. doi: 10.1056/NEJMoa1200111. Epub 2012 Mar 26. PMID 22449317
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Background] Pickard AS, De Leon MC, Kohlmann T, Cella D, Rosenbloom S. Psychometric comparison of the standard EQ-5D to a 5 level version in cancer patients. Med Care. 2007 Mar;45(3):259-63. doi: 10.1097/01.mlr.0000254515.63841.81. PMID 17304084
- [Background] Ransom D, Ashton K, Windover A, Heinberg L. Internal consistency and validity assessment of SCL-90-R for bariatric surgery candidates. Surg Obes Relat Dis. 2010 Nov-Dec;6(6):622-7. doi: 10.1016/j.soard.2010.02.039. Epub 2010 Feb 23. PMID 20627709
- [Background] Schofield CJ, Sutherland C. Disordered insulin secretion in the development of insulin resistance and Type 2 diabetes. Diabet Med. 2012 Aug;29(8):972-9. doi: 10.1111/j.1464-5491.2012.03655.x. PMID 22443306
- [Background] Sobutay E, Bilgic C, Uymaz DS, Sahin B, Mercan S, Kabaoglu B, Yapici Eser H, Yavuz Y. Can We Benefit from the Preoperative Psychometric Test with Symptom Checklist-90-Revised (SCL-90-R) to Predict Weight Loss After Sleeve Gastrectomy? Obes Surg. 2022 May;32(5):1531-1538. doi: 10.1007/s11695-022-05951-y. Epub 2022 Feb 11. PMID 35146601
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Wang Y, Beydoun MA, Liang L, Caballero B, Kumanyika SK. Will all Americans become overweight or obese? estimating the progression and cost of the US obesity epidemic. Obesity (Silver Spring). 2008 Oct;16(10):2323-30. doi: 10.1038/oby.2008.351. Epub 2008 Jul 24. PMID 18719634
- [Background] Welch GW, Jacobson AM, Polonsky WH. The Problem Areas in Diabetes Scale. An evaluation of its clinical utility. Diabetes Care. 1997 May;20(5):760-6. doi: 10.2337/diacare.20.5.760. PMID 9135939
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A; American College of Sports Medicine; American Heart Association. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1081-93. doi: 10.1161/CIRCULATIONAHA.107.185649. Epub 2007 Aug 1. PMID 17671237
- [Background] Koepsell TD, Littman AJ, Forsberg CW. Obesity, overweight, and their life course trajectories in veterans and non-veterans. Obesity (Silver Spring). 2012 Feb;20(2):434-9. doi: 10.1038/oby.2011.2. Epub 2011 Feb 3. PMID 21293452
- See also: SCL-90-R Questionnaire — https://www.pearsonassessments.com/store/usassessments/en/Store/Professional-Assessments/Personality-%26-Biopsychosocial/Symptom-Checklist-90-Revised/p/100000645.html